CLINICAL TRIAL: NCT02438787
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Study Evaluating the Efficacy and Safety of Ustekinumab in the Treatment of Anti-TNF(Alpha) Refractory Subjects With Active Radiographic Axial Spondyloarthritis
Brief Title: A Study to Evaluate the Efficacy and Safety of Ustekinumab in the Treatment of Anti-TNF(Alpha) Refractory Participants With Active Radiographic Axial Spondyloarthritis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was stopped because ustekinumab did not achieve key endpoints in a related study. The safety profile was consistent with past ustekinumab studies.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR107099; CNTO1275AKS3002 (Other: Janssen Research & Development, LLC); 2015-000288-16 (EudraCT Number)
Record Dates: First submitted 2015-05-06; First posted 2015-05-08 (Estimated); Results first posted 2018-10-01 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Axial Spondyloarthritis
Keywords: Ankylosing Spondylitis; Ustekinumab; Golimumab; STELARA
MeSH Terms: conditions — Axial Spondyloarthritis; Spondylitis, Ankylosing | interventions — Ustekinumab; golimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (placebo) (Placebo Comparator): Placebo subcutaneous (SC) injection at Weeks 0, 4, and 16. At Week 24 all participants (with the exception of participants who qualified for early escape [EE]) will be re-randomized to receive either ustekinumab 45 or 90 milligram (mg) SC injection at Weeks 24 and 28 followed by every 12 weeks (q12w) dosing, with the last administration of study agent at Week 52. Participants who meet EE criteria (less than [<] 10 percent [%] improvement from baseline in both total back pain and morning stiffness measures at both Week 12 and Week 16) will be administered open-label golimumab 50 mg SC administrations at Week 16 and every 4 weeks (q4w) thereafter through Week 52.
  Interventions: Drug: Placebo; Drug: Ustekinumab 45 mg; Drug: Ustekinumab 90 mg; Drug: Golimumab 50 mg
- Group 2 (ustekinumab 45 mg) (Experimental): Ustekinumab 45 mg SC injection at Weeks 0 and 4, followed by q12w dosing, with the last administration of study agent at Week 52. At Week 24, participants will receive placebo SC injection to maintain the blind. Participants who meet EE criteria (<10% improvement from baseline in both total back pain and morning stiffness measures at both Week 12 and Week 16) will be administered open-label golimumab 50 mg SC administrations at Week 16 and q4w thereafter through Week 52.
  Interventions: Drug: Ustekinumab 45 mg; Drug: Golimumab 50 mg
- Group 3 (ustekinumab 90 mg) (Experimental): Ustekinumab 90 mg SC injection at Weeks 0 and 4, followed by q12w dosing, with the last administration of study agent at Week 52. At Week 24, participants will receive placebo SC injection to maintain the blind. Participants who meet EE criteria (<10% improvement from baseline in both total back pain and morning stiffness measures at both Week 12 and Week 16) will be administered open-label golimumab 50 mg SC administrations at Week 16 and q4w thereafter through Week 52.
  Interventions: Drug: Ustekinumab 90 mg; Drug: Golimumab 50 mg

INTERVENTIONS:
Drug: Placebo — Placebo subcutaneous (SC) injection at Weeks 0, 4, and 16 in Group 1.
  Arms: Group 1 (placebo)
Drug: Ustekinumab 45 mg — Ustekinumab 45 mg SC injection at Weeks 24 and 28 followed by every 12 weeks (q12w) dosing, with the last administration of study agent at Week 52 in Group 1. Participants will start with ustekinumab 45 mg SC injection at Weeks 0 and 4, followed by q12w dosing, with the last administration of study agent at Week 52 in Group 2.
  Arms: Group 1 (placebo); Group 2 (ustekinumab 45 mg)
Drug: Ustekinumab 90 mg — Ustekinumab 90 mg SC injection at Weeks 24 and 28 followed by q12w dosing, with the last administration of study agent at Week 52 in Group 1. Participants will start with ustekinumab 90 mg SC injection at Weeks 0 and 4, followed by q12w dosing, with the last administration of study agent at Week 52 in Group 3.
  Arms: Group 1 (placebo); Group 3 (ustekinumab 90 mg)
Drug: Golimumab 50 mg — Participants who meet EE criteria (less than [<] 10 percent [%] improvement from baseline in both total back pain and morning stiffness measures at both Week 12 and Week 16) will be administered open-label golimumab 50 mg SC administrations at Week 16 and every 4 weeks (q4w) thereafter through Week 52 in Group 1, 2 and 3.

SUMMARY:
The purpose of this study is to assess the efficacy of ustekinumab, in adult anti-TNF(alpha) refractory participants with active radiographic axial spondyloarthritis (AxSpA), as measured by the reduction in signs and symptoms of radiographic AxSpA.

DETAILED DESCRIPTION:
This is a Phase 3, multicenter (when more than one hospital or medical school team work on a medical research study), randomized (study medication assigned to participants by chance), double-blind (neither the researchers nor the participants know what treatment the participant is receiving), placebo-controlled (an inactive substance; a pretend treatment [with no drug in it] that is compared in a clinical trial with a drug to test if the drug has a real effect) study. The study consists of 3 phases; Screening (up to 8 weeks), Treatment phase: placebo-controlled (Week 0 to 24) and active treatment (Week 24 to Week 52), and Safety Follow-up (up to 12 weeks). Participants will be randomly assigned to 1 of 3 treatment groups: placebo, ustekinumab 45 mg and ustekinumab 90 mg. The total duration of study will be up to 64 weeks. Participants will be primarily assessed for Assessment of SpondyloArthritis International Society (ASAS) 40 response at Week 24. Participants' safety will be monitored throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of definite ankylosing spondylitis (AS), as defined by the modified 1984 New York criteria. The radiographic criterion must be confirmed by a central xray reader and at least 1 clinical criterion must be met
* Participants must have symptoms of active disease at screening and at baseline, as evidenced by both a Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score of greater than or equal to (>=4) and a visual analog scale (VAS) score for total back pain of >=4, each on a scale of 0 to 10
* Participants with elevated high sensitivity C-reactive protein (hsCRP) level of >=0.300 milligram per deciliter (mg/dL) at screening
* Refractory by either lack of benefit or documented intolerance to 1 and no more than 1 anti-TNF(alpha) agent
* Inadequate response to at least 2 nonsteroidal anti-inflammatory drugs (NSAIDs) over a 4-week period in total with maximal doses of NSAID(s), or is unable to receive a full 4 weeks of maximal NSAID therapy because of intolerance, toxicity, or contraindications to NSAIDs.
* Participants with complete ankylosis of the spine are permitted to be included in the study, but will be limited to approximately 10 percent (%) of the study population

Exclusion Criteria:

* Participants who have other inflammatory diseases that might confound the evaluations of benefit from the ustekinumab therapy, including but not limited to, rheumatoid arthritis, systemic lupus erythematosus, or Lyme disease
* Participants who have received infliximab or infliximab biosimilar, within 12 weeks of the first study agent administration; have received adalimumab, adalimumab biosimilar, or certolizumab pegol within 6 weeks of the first study agent administration; have received etanercept or etanercept biosimilar within 6 weeks of the first study agent administration
* Participants who have ever received golimumab
* Participants who are pregnant, nursing, or planning a pregnancy or fathering a child while enrolled in the study or within 5 months after receiving the last administration of study agent
* Participants who have received any systemic immunosuppressives or disease-modifying antirheumatic drugs (DMARDs) other than methotrexate (MTX), sulfasalazine (SSZ), or hydroxychloroquine (HCQ) within 4 weeks prior to first administration of study agent. Medications in these categories include, but are not limited to leflunomide, chloroquine, azathioprine, cyclosporine, mycophenolate mofetil, gold, and penicillamine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2015-07-31 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (148):
- United States (19):
  - Glendale, Arizona
  - Peoria, Arizona
  - Phoenix, Arizona
  - Fremont, California
  - St. Petersburg, Florida
  - Tampa, Florida
  - Boise, Idaho
  - Chicago, Illinois
  - Monroe, Louisiana
  - Eagan, Minnesota
  - Orchard Park, New York
  - Portland, Oregon
  - Duncansville, Pennsylvania
  - Wyomissing, Pennsylvania
  - Jackson, Tennessee
  - Austin, Texas
  - Mesquite, Texas
  - Arlington, Virginia
  - Seattle, Washington
- Argentina (5):
  - Buenos Aires
  - Ciudad de Buenos Aires
  - Ciudad de La Plata
  - Ciudad de San Miguel de Tucuman
  - Córdoba
- Belgium (6):
  - Brussels
  - Genk
  - Ghent
  - Leuven
  - Liège
  - Merksem (Antwerp)
- Brazil (8):
  - Campinas
  - Curitiba
  - Goiânia
  - Juiz de Fora
  - Porto Alegre
  - Rio de Janeiro
  - Santo André
  - São Paulo
- Bulgaria (5):
  - Burgas
  - Pleven
  - Plovdiv
  - Rousse
  - Sofia
- Canada (5):
  - Victoria, British Columbia
  - St. John's, Newfoundland and Labrador
  - Toronto, Ontario
  - Windsor, Ontario
  - Québec, Quebec
- Czechia (5):
  - Bruntál
  - Pardubice
  - Prague
  - Uherské Hradiště
  - Zlín
- France (8):
  - Boulogne-Billancourt
  - Chambray-lès-Tours
  - Échirolles
  - Montpellier
  - Orléans
  - Paris
  - Rouen
  - Toulouse
- Germany (8):
  - Bad Neuheim
  - Berlin
  - Cologne
  - Gommern
  - Hamburg
  - Herne
  - Olsberg
  - Ratingen
- Hungary (8):
  - Budapest
  - Debrecen
  - Eger
  - Kistarcsa
  - Nyíregyháza
  - Székesfehérvár
  - Szolnok
  - Veszprém
- Mexico (3):
  - Culiacán
  - Guadalajara
  - Mexico City
- Poland (7):
  - Bialystok
  - Bydgoszcz
  - Elblag
  - Nadarzyn
  - Szczecin
  - Torun
  - Warsaw
- Portugal (3):
  - Almada
  - Lisbon
  - Porto
- Russia (17):
  - Belgorod
  - Chelyabinsk
  - Chita
  - Kazan'
  - Kemerovo
  - Khanty-Mansiysk
  - Kursk
  - Moscow
  - Nizhny Novgorod
  - Omsk
  - Orenburg
  - Petrozavodsk
  - Pyatigorsk
  - Saint Petersburg
  - Saratov
  - Ufa
  - Zelenograd
- South Korea (6):
  - Daegu
  - Daejeon
  - Gwangju
  - Jeonju
  - Seoul
  - Suwon
- Spain (11):
  - A Coruña
  - Barcelona
  - Bilbao
  - Córdoba
  - L'Hospitalet de Llobregat
  - Madrid
  - Málaga
  - Sabadell
  - Santiago de Compostela
  - Seville
  - Valencia
- Taiwan (7):
  - Changhua
  - Hualien City
  - Kaohsiung City
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan District
- Ukraine (11):
  - Cherkasy
  - Ivano-Frankivsk
  - Kharkiv
  - Kyiv
  - Lviv
  - Odesa
  - Poltava
  - Ternopil
  - Uzhhorod
  - Vinnytsia
  - Zaporizhzhya
- United Kingdom (6):
  - Bath
  - Leytonstone
  - London
  - Peterborough
  - Stoke-on-Trent
  - Upton

REFERENCES:
- [Derived] Kavanaugh A, Baraliakos X, Gao S, Chen W, Sweet K, Chakravarty SD, Song Q, Shawi M, Rahman P. Genetic and Molecular Distinctions Between Axial Psoriatic Arthritis and Radiographic Axial Spondyloarthritis: Post Hoc Analyses from Four Phase 3 Clinical Trials. Adv Ther. 2023 May;40(5):2439-2456. doi: 10.1007/s12325-023-02475-4. Epub 2023 Mar 30. PMID 36995469
- [Derived] Deodhar A, Gensler LS, Sieper J, Clark M, Calderon C, Wang Y, Zhou Y, Leu JH, Campbell K, Sweet K, Harrison DD, Hsia EC, van der Heijde D. Three Multicenter, Randomized, Double-Blind, Placebo-Controlled Studies Evaluating the Efficacy and Safety of Ustekinumab in Axial Spondyloarthritis. Arthritis Rheumatol. 2019 Feb;71(2):258-270. doi: 10.1002/art.40728. Epub 2018 Dec 29. PMID 30225992

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 315 participants were randomized and treated (104 participants to placebo, 106 participants to ustekinumab 45 milligram (mg), and 105 participants to 90 mg).
Groups:
- Placebo: Participants received placebo subcutaneous (SC) injection at Weeks 0, 4, and 16. At Week 16, participants who met early escape (EE) criteria were administered open-label golimumab 50 mg SC administrations at Week 16 and every 4 Weeks (q4w) thereafter through Week 52. At Week 24 all participants (with the exception of participants who qualified for EE) were re-randomized to receive either ustekinumab 45 or 90 mg SC injection at Weeks 24 and 28 followed by every 12 weeks (q12w) dosing, with the last administration of study agent at Week 52.
- Ustekinumab 45mg: Participants received ustekinumab 45 mg SC injection at Weeks 0 and 4, followed by q12w dosing, with the last administration of study agent at Week 52. At Week 16, participants who met EE criteria were administered open label golimumab 50 mg SC administrations at Week 16 and q4w thereafter through Week 52. At Week 24,participants were to receive placebo SC injection to maintain the blind.
- Ustekinumab 90mg: Participants received Ustekinumab 90 mg SC injection at Weeks 0 and 4, followed by q12w dosing, with the last administration of study agent at Week 52. At Week 16, participants who met EE criteria were administered open label golimumab 50 mg SC administrations at Week 16 and q4w thereafter through Week 52. At Week 24,participants were to receive placebo SC injection to maintain the blind.
Period: Overall Study
Arm/Group | Placebo | Ustekinumab 45mg | Ustekinumab 90mg
Started | 104 | 106 | 105
Early Escape at Week 16 | 21 (Study discontinuation/completion reported under randomization group) | 21 (Study discontinuation/completion reported under randomization group) | 20 (Study discontinuation/completion reported under randomization group)
Cross Over at Week 24 | 43 (Out of 43: crossed over to Ustekinumab 45 mg (n=21) and Ustekinumab 90 mg (n=22)) | 0 | 0
Completed | 23 | 23 | 22
Not Completed | 81 | 83 | 83
Not completed — Adverse Event | 1 | 0 | 2
Not completed — Lack of Efficacy | 1 | 2 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 15 | 7 | 10
Not completed — Study discontinued by sponsor | 64 | 72 | 69
Not completed — Other | 0 | 1 | 0
Not completed — Site terminated by sponsor | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) includes all participants who were randomized and received at least one administration of study agent.
Groups:
- Placebo: Participants received placebo SC injection at Weeks 0, 4, and 16. At Week 16, participants who met EE criteria were administered open-label golimumab 50 mg SC administrations at Week 16 and q4w thereafter through Week 52. At Week 24 all participants (with the exception of participants who qualified for EE) were re-randomized to receive either ustekinumab 45 or 90 mg SC injection at Weeks 24 and 28 followed by every 12 weeks (q12w) dosing, with the last administration of study agent at Week 52.
- Ustekinumab 45mg: Participants received ustekinumab 45 mg SC injection at Weeks 0 and 4, followed by q12w dosing, with the last administration of study agent at Week 52. At Week 16, participants who met EE criteria were administered open-label golimumab 50 mg SC administrations at Week 16 and q4w thereafter through Week 52. At Week 24,participants were to receive placebo SC injection to maintain the blind.
- Ustekinumab 90mg: Participants received Ustekinumab 90 mg SC injection at Weeks 0 and 4, followed by q12w dosing, with the last administration of study agent at Week 52. At Week 16, participants who met EE criteria were administered open-label golimumab 50 mg SC administrations at Week 16 and q4w thereafter through Week 52. At Week 24,participants were to receive placebo SC injection to maintain the blind.
- Total: Total of all reporting groups
Arm/Group | Placebo | Ustekinumab 45mg | Ustekinumab 90mg | Total
Number analyzed (Participants) | 104 | 106 | 105 | 315
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.8 (11.72) | 41.4 (11.33) | 41.5 (11.02) | 41.2 (11.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 18 | 13 | 55
  Male | 80 | 88 | 92 | 260
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 14 | 16 | 42
  Not Hispanic or Latino | 91 | 91 | 88 | 270
  Unknown or Not Reported | 1 | 1 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 14 | 16 | 14 | 44
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2
  White | 82 | 84 | 84 | 250
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 7 | 5 | 7 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 14 | 16 | 14 | 44
  Black or African American | 1 | 1 | 0 | 2
  Hispanic or Latino | 4 | 8 | 10 | 22
  Other | 8 | 6 | 8 | 22
  White Non-Hispanic | 77 | 75 | 73 | 225
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 2 | 3 | 2 | 7
  BELGIUM | 3 | 1 | 1 | 5
  BRAZIL | 3 | 2 | 5 | 10
  BULGARIA | 5 | 3 | 5 | 13
  CANADA | 1 | 0 | 1 | 2
  CZECH REPUBLIC | 1 | 1 | 1 | 3
  FRANCE | 0 | 1 | 1 | 2
  GERMANY | 2 | 4 | 3 | 9
  HUNGARY | 4 | 9 | 6 | 19
  MEXICO | 8 | 7 | 7 | 22
  POLAND | 5 | 5 | 5 | 15
  PORTUGAL | 1 | 0 | 0 | 1
  RUSSIAN FEDERATION | 19 | 27 | 23 | 69
  SOUTH KOREA | 6 | 5 | 3 | 14
  SPAIN | 3 | 4 | 4 | 11
  TAIWAN | 8 | 10 | 11 | 29
  UKRAINE | 28 | 16 | 22 | 66
  UNITED KINGDOM | 3 | 4 | 3 | 10
  UNITED STATES | 2 | 4 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved an Assessment of SpondyloArthritis International Society (ASAS) 40 Response at Week 24
Description: ASAS 40 defined as improvement from baseline of greater than or equal to (>=) 40% and with an absolute improvement from baseline of at least 2 on 0 to10cm scale in at least 3 of following 4 domains: Patient's global assessment (0 to 10cm; 0=very well,10=very poor),total back pain (0 to 10cm; 0=no pain,10=most severe pain), BASFI(self-assessment represented as mean (0 to 10 cm; 0=easy to 10=impossible) of 10 questions, 8 of which relate to participant's functional anatomy and 2 relate to participant's ability to cope with everyday life), Inflammation (0 to 10cm;0=none,10=very severe); no worsening at all from baseline in remaining domain. ASAS40 response based on imputed data using treatment failure(consider non-responders at and after treatment failure),early escape rules(consider non-responder at Week 20 and 24),non-responder[NRI(non responder imputation)] (missing responses at post baseline visit imputed as non-responder).
Time Frame: Week(W) 24
Population: Modified-FAS included FAS population, excluding who discontinued study agent prior to W24 due to trial termination,not had efficacy assessments at W24,but not excluding participants who met EE at W16/ had treatment failure prior to W24.Participants analyzed based on randomized treatment group they were assigned to regardless of treatment received.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab 45mg | Ustekinumab 90mg
Number analyzed (Participants) | 73 | 73 | 67
Percentage of participants | 12.3 | 19.2 | 26.9

2. Secondary Outcome: Percentage of Participants Who Achieved an ASAS 20 Response at Week 24
Description: ASAS 20 defined as improvement from baseline of >= 20% from baseline and with an absolute improvement from baseline of 1 on a 0 to 10 cm scale in at least 3 of following 4 domains: Patient's global assessment (0 to 10cm; 0=very well,10=very poor),total back pain (0 to 10cm; 0=no pain,10=most severe pain), BASFI (self-assessment represented as mean (0 to 10 cm; 0=easy to 10=impossible) of 10 questions, 8 of which relate to participant's functional anatomy and 2 relate to participant's ability to cope with everyday life), Inflammation (0 to 10cm;0=none,10=very severe); absence of deterioration (>= 20% and worsening of at least 1 on a 0 to 10 cm scale) from baseline in the potential remaining domain. ASAS20 response based on imputed data using treatment failure(consider non-responders at and after treatment failure),early escape rules(consider non-responder at Week 20 and 24),non-responder[NRI] (missing responses at post baseline visit imputed as non-responder).
Time Frame: Week 24
Population: Modified-FAS population was used. Participants analyzed based on randomized treatment group they were assigned to regardless of treatment received.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab 45mg | Ustekinumab 90mg
Number analyzed (Participants) | 73 | 73 | 67
Percentage of participants | 27.4 | 31.5 | 37.3

3. Secondary Outcome: Percentage of Participants Who Achieved at Least a 50 Percent (%) Improvement From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at Week 24
Description: BASDAI is used to measure the ankylosing spondylitis (AS) disease severity. It consists of 6 questions: fatigue, spinal pain, arthralgia (joint pain) or swelling, enthesitis (inflammation of tendons and ligaments), morning stiffness(MS) (2 questions: duration and severity). Each question is an easy to answer 10 cm visual analog scale (VAS), with 0 being none, and 10 being very severe and for the last question related to MS duration: 0(0 hours), 10(2 or more hours). In order to give each of 5 symptoms equal weight, mean of 2 questions about MS will be added to total of remaining 4 scores, final BASDAI score (ranging 0-10) is average of overall total score. Higher BASDAI score indicates more severe AS symptom. 50% improvement in response based on imputed data using treatment failure(consider non-responders at and after treatment failure),early escape rules(consider non-responder at Week 20 and 24),non-responder[NRI] (missing responses at post baseline visit imputed as non-responder).
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab 45mg | Ustekinumab 90mg
Number analyzed (Participants) | 73 | 73 | 67
Percentage of participants | 11.0 | 15.1 | 28.4

4. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) Total Score at Week 24
Description: The BASFI is composed with 10 questions (each question is answered with a visual analogue scale 0-10 cm) to assess the disease severity, including the first 8 questions regarding to functional anatomy related activities and the remaining 2 questions related to daily activities of AS participants. Each question is a 10cm VAS with a value between 0 (easy) and 10 (impossible). The final BASFI score is the mean of the 10 scores. The BASFI score is the average of the 10 responses and has a possible minimum value of 0 and a possible maximum value of 10. Higher BASFI score indicates more severe functional limitations of the participant due to AS. Missing data were imputed using early escape rule (consider non-responder at Week 20 and 24).
Time Frame: Baseline and Week 24
Population: Modified-FAS population was used. Participants analyzed based on randomized treatment group they were assigned to regardless of treatment received. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this endpoint.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ustekinumab 45mg | Ustekinumab 90mg
Number analyzed (Participants) | 44 | 44 | 42
Units on a scale | -1.29 (2.219) | -1.74 (2.724) | -2.17 (2.438)

5. Secondary Outcome: Percentage of Participants Who Achieved Ankylosing Spondylitis Disease Activity Score-C Reactive Protein (ASDAS-CRP) Inactive Disease (<1.3) at Week 24
Description: ASDAS includes CRP mg/L; four additional self-reported items (rated on 0-10cm VAS or 0-10 numerical rating scale [NRS]) included are total back pain (TBP), duration of morning stiffness (DMS), peripheral pain/swelling and patient global assessment (PGA). ASDAS scores calculated as: ASDAS(CRP) = (0.121*total back pain) + (0.110*participant global) + (0.073*peripheral pain/swelling) + (0.058* duration of morning stiffness) + (0.579*Ln(CRP+1). The disease activity, TBP, and peripheral pain/swelling on a numeric rating scale (from 0 (normal) to 10 (very severe)) and DMS on a numeric rating scale (0 to 10, with 0 being none and 10 representing a duration of =>2 hours). Inactive disease is defined as an ASDAS score <1.3. ASDAS (CRP) Inactive Disease is based on imputed data using treatment failure(consider non-responders at and after treatment failure),early escape rules(consider non-responder at Week 20 and 24), NRI(missing responses at post baseline visit imputed as non-responder).
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab 45mg | Ustekinumab 90mg
Number analyzed (Participants) | 73 | 73 | 67
Percentage of participants | 0 | 2.7 | 3.0

6. Secondary Outcome: Change From Baseline in High Sensitivity C-Reactive Protein (hsCRP) Levels Through Week 24
Description: Change from baseline in hsCRP was reported. hsCRP is a sensitive laboratory assay for serum levels of C-Reactive Protein, which is a biomarker of inflammation. Early escape rule was applied (measurement value at Week 20 and Week 24 was set as missing).
Time Frame: Baseline, Week 4, 8, 12, 16, 20 and 24
Population: Modified-FAS population was used. Participants analyzed based on randomized treatment group they were assigned to regardless of treatment received. Here 'n' signifies number of participants analyzed for this endpoint at specific timepoints.
Measure: Mean (Standard Deviation); unit: Milligrams per deciliter (mg/dL)
Arm/Group | Placebo | Ustekinumab 45mg | Ustekinumab 90mg
Number analyzed (Participants) | 73 | 73 | 67
Milligrams per deciliter (mg/dL)
  Change at Week 4: number analyzed (Participants) | 71 | 69 | 67
  Change at Week 4 | 0.12 (2.211) | -0.35 (2.171) | -0.12 (1.604)
  Change at Week 8: number analyzed (Participants) | 69 | 68 | 65
  Change at Week 8 | -0.18 (2.526) | -0.54 (2.213) | -0.24 (2.555)
  Change at Week 12: number analyzed (Participants) | 68 | 68 | 64
  Change at Week 12 | -0.02 (2.836) | -0.36 (2.495) | 0.05 (2.842)
  Change at Week 16: number analyzed (Participants) | 66 | 67 | 64
  Change at Week 16 | -0.06 (2.676) | -0.21 (2.333) | 0.12 (2.720)
  Change at Week 20: number analyzed (Participants) | 42 | 45 | 44
  Change at Week 20 | 0.23 (2.266) | -0.11 (1.611) | -0.40 (2.198)
  Change at Week 24: number analyzed (Participants) | 43 | 44 | 43
  Change at Week 24 | -0.36 (2.067) | -0.14 (2.041) | -0.26 (1.850)

7. Secondary Outcome: Percentage of Participants With ASDAS (CRP) Inactive Disease (<1.3) at Week 4, 8, 12, 16 and 20
Description: ASDAS includes CRP mg/L; four additional self-reported items (rated on 0-10cm VAS or 0-10 numerical rating scale [NRS]) included are total back pain (TBP), duration of morning stiffness (DMS), peripheral pain/swelling and patient global assessment (PGA). ASDAS scores calculated as: ASDAS(CRP) = (0.121*total back pain) + (0.110*participant global) + (0.073*peripheral pain/swelling) + (0.058* duration of morning stiffness) + (0.579*Ln(CRP+1)). The disease activity, TBP, and peripheral pain/swelling on a numeric rating scale (from 0 (normal) to 10 (very severe) and DMS on a numeric rating scale (0 to 10, with 0 being none and 10 representing a duration of =>2 hours). Inactive disease is defined as an ASDAS score <1.3. ASDAS (CRP) Inactive Disease is based on imputed data using treatment failure(consider non-responders at and after treatment failure),early escape rules(consider non-responder at Week 20 and 24), NRI(missing responses at post baseline visit imputed as non- responders).
Time Frame: Week 4, 8, 12, 16 and 20
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab 45mg | Ustekinumab 90mg
Number analyzed (Participants) | 73 | 73 | 67
Percentage of participants
  Week 4 | 0 | 0 | 0
  Week 8 | 0 | 2.7 | 0
  Week 12 | 0 | 1.4 | 3.0
  Week 16 | 0 | 1.4 | 3.0
  Week 20 | 1.4 | 1.4 | 1.5

8. Secondary Outcome: Percentage of Participants Who Achieved ASAS 40 Responses at Week 4, 8, 12, 16 and 20
Description: ASAS 40 defined as improvement from baseline >= 40% and with an absolute improvement from baseline of at least 2 on 0 to10cm scale in at least 3 of following 4 domains: Patient's global assessment (0 to 10cm; 0=very well,10=very poor),total back pain (0 to 10cm; 0=no pain,10=most severe pain), BASFI (self-assessment represented as mean (0 to 10 cm; 0=easy to 10=impossible) of 10 questions, 8 of which relate to participant's functional anatomy and 2 relate to participant's ability to cope with everyday life), Inflammation (0 to 10cm;0=none,10=very severe); no worsening at all from baseline in remaining domain. ASAS40 response based on imputed data using treatment failure(consider non-responders at and after treatment failure),early escape rules(consider non-responder at Week 20 and 24),non-responder[NRI] (missing responses at post baseline visit imputed as non-responder).
Time Frame: Week 4, 8, 12, 16 and 20
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab 45mg | Ustekinumab 90mg
Number analyzed (Participants) | 73 | 73 | 67
Percentage of participants
  Week 4 | 6.8 | 8.2 | 11.9
  Week 8 | 11.0 | 12.3 | 16.4
  Week 12 | 6.8 | 15.1 | 19.4
  Week 16 | 9.6 | 15.1 | 20.9
  Week 20 | 12.3 | 21.9 | 25.4

9. Secondary Outcome: Percentage of Participants Who Achieved ASAS 20 Responses at Week 4, 8, 12, 16 and 20
Description: ASAS 20 defined as improvement from baseline of >= 20% and with an absolute improvement from baseline of 1 on a 0 to 10 cm scale in at least 3 of following 4 domains: Patient's global assessment (0 to 10cm; 0=very well,10=very poor),total back pain (0 to 10cm; 0=no pain,10=most severe pain), BASFI (self-assessment represented as mean (0 to 10 cm; 0=easy to 10=impossible) of 10 questions, 8 of which relate to participant's functional anatomy and 2 relate to participant's ability to cope with everyday life), Inflammation (0 to 10cm;0=none,10=very severe); absence of deterioration (>= 20% and worsening of at least 1 on a 0 to 10 cm scale) from baseline in the potential remaining domain. ASAS20 response based on imputed data using treatment failure(consider non-responders at and after treatment failure),early escape rules(consider non-responder at Week 20 and 24),non-responder[NRI] (missing responses at post baseline visit imputed as non-responder).
Time Frame: Week 4, 8, 12, 16 and 20
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab 45mg | Ustekinumab 90mg
Number analyzed (Participants) | 73 | 73 | 67
Percentage of participants
  Week 4 | 19.2 | 26.0 | 31.3
  Week 8 | 20.5 | 34.2 | 29.9
  Week 12 | 24.7 | 30.1 | 32.8
  Week 16 | 23.3 | 21.9 | 35.8
  Week 20 | 28.8 | 35.6 | 41.8

10. Secondary Outcome: Percentage of Participants Who Achieved at Least a 50% Improvement From Baseline in BASDAI at Week 4, 8, 12, 16 and 20
Description: as for outcome 3
Time Frame: Week 4, 8, 12, 16 and 20
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ustekinumab 45mg | Ustekinumab 90mg
Number analyzed (Participants) | 73 | 73 | 67
Percentage of participants
  Week 4 | 5.5 | 6.8 | 11.9
  Week 8 | 8.2 | 11.0 | 13.4
  Week 12 | 4.1 | 15.1 | 11.9
  Week 16 | 11.0 | 15.1 | 16.4
  Week 20 | 8.2 | 16.4 | 19.4

11. Secondary Outcome: Change From Baseline in BASFI Total Score at Week 4, 8, 12, 16 and 20
Description: as for outcome 4
Time Frame: Baseline, Week 4, 8, 12, 16 and 20
Population: Modified-FAS population was used. Participants analyzed based on randomized treatment group they were assigned to regardless of treatment received. Here 'n' (number analyzed) signifies number of participants who were analyzed at each specified timepoint, for each arm, respectively.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ustekinumab 45mg | Ustekinumab 90mg
Number analyzed (Participants) | 73 | 73 | 67
Units on a scale
  Change at Week 4: number analyzed (Participants) | 71 | 69 | 66
  Change at Week 4 | -0.58 (1.571) | -0.69 (1.662) | -0.73 (1.915)
  Change at Week 8: number analyzed (Participants) | 69 | 68 | 64
  Change at Week 8 | -0.66 (2.099) | -0.86 (2.010) | -1.02 (2.010)
  Change at Week 12: number analyzed (Participants) | 68 | 68 | 63
  Change at Week 12 | -0.73 (2.406) | -0.70 (2.380) | -0.77 (2.459)
  Change at Week 16: number analyzed (Participants) | 66 | 67 | 63
  Change at Week 16 | -0.58 (2.053) | -0.54 (2.491) | -0.80 (2.574)
  Change at Week 20: number analyzed (Participants) | 41 | 45 | 43
  Change at Week 20 | -1.45 (2.353) | -1.73 (2.564) | -2.16 (2.140)

ADVERSE EVENTS:
Time Frame: Up to Week 64
Description: The safety analysis set included all participants who received at least 1 (partial or complete) administration of study agent, i.e., the treated population. Adverse events were reported according to the treatment they actually received, regardless of the treatments they are randomized to.
Groups:
- Placebo: Participants received placebo SC injection at Weeks 0, 4, and 16. At Week 16, participants who met EE criteria were administered open-label golimumab 50 mg SC administrations at Week 16 and q4w thereafter through Week 52. At Week 24 all participants (with the exception of participants who qualified for EE) were re-randomized to receive either ustekinumab 45 or 90 mg SC injection at Weeks 24 and 28 followed by every 12 weeks (q12w) dosing. Included all participants, but adverse events for participants who early escaped at Week 16 or crossed over at Week 24 are only counted up to Week 16 or Week 24 respectively.
- Placebo to Golimumab: Participants randomized to placebo SC who met early escape criteria and received golimumab from Week 16; adverse events are counted from early escape onward.
- Placebo to Ustekinumab 45mg: Participants randomized to placebo SC and then rerandomized to receive ustekinumab 45 mg at Week 24; adverse events are counted from crossover onward.
- Placebo to Ustekinumab 90mg: Participants randomized to placebo SC and then rerandomized to receive ustekinumab 90 mg at Week 24; adverse events are counted from crossover onward.
- Ustekinumab 45mg Only: Participants received ustekinumab 45 mg SC injection at Weeks 0 and 4, followed by q12w dosing. Adverse events for participants who early escaped at Week 16 are only counted up to Week 16.
- Ustekinumab 45mg to Golimumab: Participants randomized to ustekinumab 45 mg SC who met early escape criteria and received golimumab from Week 16; adverse events are counted from early escape onward.
- Ustekinumab 90mg Only: Participants received Ustekinumab 90 mg SC injection at Weeks 0 and 4, followed by q12w dosing. Adverse events for participants who early escaped at Week 16 are only counted up to Week 16.
- Ustekinumab 90mg to Golimumab: Participants randomized to ustekinumab 90 mg SC who met early escape criteria and received golimumab from Week 16; adverse events are counted from early escape onward.
Arm/Group | Placebo | Placebo to Golimumab | Placebo to Ustekinumab 45mg | Placebo to Ustekinumab 90mg | Ustekinumab 45mg Only | Ustekinumab 45mg to Golimumab | Ustekinumab 90mg Only | Ustekinumab 90mg to Golimumab
All-Cause Mortality (participants affected / at risk) | 0/104 | 0/21 | 0/21 | 0/22 | 0/106 | 0/21 | 0/105 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/104 | 2/21 | 0/21 | 1/22 | 3/106 | 1/21 | 6/105 | 1/20
Other Adverse Events (participants affected / at risk) | 19/104 | 0/21 | 2/21 | 1/22 | 19/106 | 7/21 | 18/105 | 10/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=104) | Placebo to Golimumab (N=21) | Placebo to Ustekinumab 45mg (N=21) | Placebo to Ustekinumab 90mg (N=22) | Ustekinumab 45mg Only (N=106) | Ustekinumab 45mg to Golimumab (N=21) | Ustekinumab 90mg Only (N=105) | Ustekinumab 90mg to Golimumab (N=20)
Myocardial Ischaemia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Iritis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Axial Spondyloarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal Amyloidosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Uterine Polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Uterine Prolapse (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=104) | Placebo to Golimumab (N=21) | Placebo to Ustekinumab 45mg (N=21) | Placebo to Ustekinumab 90mg (N=22) | Ustekinumab 45mg Only (N=106) | Ustekinumab 45mg to Golimumab (N=21) | Ustekinumab 90mg Only (N=105) | Ustekinumab 90mg to Golimumab (N=20)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 4 | 1 | 1 | 1
Vitreous Haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mouth Ulceration (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Injection Site Bruising (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 2 | 0 | 0 | 0 | 3 | 0 | 1 | 1
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Viral Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 4 | 0 | 0 | 0 | 4 | 2 | 8 | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Alanine Aminotransferase Increased (Investigations) | 6 | 0 | 0 | 1 | 2 | 2 | 4 | 2
Aspartate Aminotransferase Increased (Investigations) | 5 | 0 | 0 | 1 | 2 | 2 | 3 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Skin Disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The study was discontinued before it was fully enrolled due to lack of efficacy of either dose of ustekinumab in the CNTO1275AKS3001 (NCT02437162) study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2015-07-13): https://cdn.clinicaltrials.gov/large-docs/87/NCT02438787/Prot_001.pdf
  • Statistical Analysis Plan (2017-04-14): https://cdn.clinicaltrials.gov/large-docs/87/NCT02438787/SAP_000.pdf